CLINICAL TRIAL: NCT06056492
Title: Effectiveness of Children Experiencing Nitrous Oxide/Oxygen Inhalation Sedation at an Assessment Visit Before Having Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Richard Balmer (Other)
Responsible Party: Sponsor-Investigator, Dr Richard Balmer, Associate Professor Paediatric Dentistry, University of Leeds
Organization: University of Leeds (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULeeds1
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants assigned to the control group received assessment without experience N2O/O2 sedation and they tried the mask with O2 only.
  Interventions: Behavioral: Experience of nitrous oxide sedation at assessment
- Study Group (Experimental): Participants assigned to the study group received assessment with experience of N2O/O2 sedation
  Interventions: Behavioral: Experience of nitrous oxide sedation at assessment

INTERVENTIONS:
Behavioral: Experience of nitrous oxide sedation at assessment — Apart from the Lead researcher, a dental nurse assisted with the dental treatment on every appointment. A specially trained sedation nurse was responsible for the monitoring during sedation. The Porter Brown inhalation sedation machine (RA Services, Keighly, W. Yorkshire, UK) was used. Once the appropriate nasal hood was selected, 100% O2 was introduced for 1-2 minutes. Following that, the level of N2O was increased in 10% increments until signs of sedation were observed. The endpoint was between 30-40% nitrous oxide.

SUMMARY:
The purpose of this study is to find out the effect of experience of dental sedation at assessment on children's anxiety before the actual treatment session.

DETAILED DESCRIPTION:
Title: Effectiveness of children experiencing nitrous oxide/oxygen inhalation sedation at an assessment visit before having treatment.

Background: Dental anxiety is a common problem, affecting people of all ages, but predominantly children and adolescents. Inhalation sedation (IHS) using nitrous oxide/oxygen (N2O/O2) mixture is a pharmacological behaviour management technique that is widely used to manage dental anxiety in children. It is suggested that the use of an acclimatisation would increase the acceptability and the efficacy of N2O/O2 success. Even though the introductory appointment has been widely proposed, there have not been any studies conducted to measure the effectiveness of this appointment in improving the success of N2O/O2 sedation in children.

Aims: This study aimed to investigate the effect of experience of nitrous oxide/oxygen sedation at assessment prior to dental inhalation sedation on children's anxiety.

Methods: The study was a parallel randomised non blinded control clinical trial. Children aged five to fifteen years who were seen at the Leeds Dental Institute for dental treatment under inhalation sedation were recruited on the assessment appointment (1st visit). Both two groups received an assessment appointment, however participants of the study group tried on the mask and the nitrous oxide/oxygen sedation while the ones of the control group tried on the mask without the nitrous oxide/oxygen sedation. Following the assessment appointment, both groups received a second appointment for treatment. Dental anxiety was measured through two different methods. Primarily through the MCDASf questionnaire, which was completed once at the beginning of the assessment visit and twice at the beginning and end of the treatment visit. Secondarily anxiety was measured though the E4 wristband which participants of both groups wore throughout both appointments and recorded their Heart Rate (HR) and Skin Temperature (ST). At the end of the treatment visit, participants and their parents/legal guardians were asked to complete a feedback questionnaire related to the E4 wristband and the experience of N2O/O2 sedation at the assessment visit.

- 6 -

ELIGIBILITY:
Inclusion Criteria:

Patients attending the Sedation Unit for dental treatment under inhalation sedation.

* Children aged 5 to 15 years.
* ASA Class I or II.
* First time having inhalation sedation.

Exclusion Criteria:

* Participants who refuse to wear the mask.

  * Language barriers where no interpreter was available
  * Parents/Carer who refused to sign consent or children who did not assent.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Modified Child Dental Anxiety Scale | At start of recruitment. 4 weeks. 4 weeks.
  Score 8-40. High score is high anxiety. Measured through MCDAS and E$ physiological wristband data

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom